CLINICAL TRIAL: NCT06871618
Title: Retrospective Study of Surgical Induced Abortions Between 14 and 16 Weeks of Amenorrhea At Croix Rousse University Hospital in Lyon
Acronym: TARDIVG
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5192
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Induced Abortion; Instrumental Induced Abortion Between 14 and 16 Weeks of Amenorrhea
Keywords: interruption of pregnancy; Induced abortion; instrumental technique; women complications
MeSH Terms: interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women who undergone a surgical induced abortion before 14AW: Women who undergone a surgical induced abortion at Croix Rousse Hospital in Lyon between March 2022 and March 2023 before 14AW
  Interventions: Other: Retrospective
- Women who undergone a surgical induced abortion between 14 and 16AW.: Women who undergone a surgical induced abortion at Croix Rousse Hospital in Lyon between March 2022 and March 2023 between 14 and 16AW.

INTERVENTIONS:
Other: Retrospective — Retrospective Operative risk in patients undergoing instrumental abortion
  Groups: Women who undergone a surgical induced abortion before 14AW

SUMMARY:
In France, induced abortions can be carried out by two different methods: the medicinal one, which involves taking medications to expel the pregnancy (MIFEPRISTONE and then MISOPROSTOL), and the instrumental one, which involves aspiration in the operating room.

According to the high authority of health, before 9 weeks of amenorrhea, both methods are possible if there is no contraindication to one of them. After 9 weeks of amenorrhea, only the instrumental method is authorized.

Until March 2022, the maximal deadline to abort was 14 weeks of amenorrhea. On March 2nd 2022, a change in the law extended this time limit from 14 to 16 weeks of amenorrhea. Only one study was carried out following this change in France to assess the complication rate of late abortions (between 14 and 16 weeks of amenorrhea (AW)). This study was carried out at Trousseau Hospital in Paris, with a total of 46 patients. The results of this study were reassuring, with bleeding > 500 mL for only one patient (2.2%, 95% CI [0.0-6.4]) and no complications such as perforation, postoperative infection or revision surgery, or need for transfusion.

However, this paper is the only French study which evaluated the operative risks of late abortion since the change in the law, and its power is small. There is a need to assess the operative risks of late abortion on a larger cohort.

That's why the investigators had the idea to conduct a study looking at all instrumental abortions performed in Croix Rousse Hospital in Lyon between March 2022 and March 2023, representing around 700 procedures. The aim of the study is to compare the complication rates of instrumental abortions between 14 and 16 weeks of amenorrhea versus those carried out before 14 weeks.

ELIGIBILITY:
Eligibility Criteria *

* Inclusion Criteria * :

  * Surgical induced abortion
  * At Croix Rousse hospital, Lyon
  * Between March 2022 and March 2023
* Exclusion Criteria * :

  * Minor patients

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Adult women who undergone a surgical abortion at Croix Rousse Hospital in Lyon between March 2022 and March 2023.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with intraoperative bleeding > 500 mL | Primary endpoint is measured during the intervention by collecting the total blood quantity collected into a reservoir connected to the aspiration probe.
  Evaluated by collecting blood loss during the procedure (in 50 mL increments)

CONTACTS AND LOCATIONS:
Locations (1):
- Croix Rousse University Hospital, Lyon, France